CLINICAL TRIAL: NCT06182696
Title: An Open Label,Multi-center Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Autologous T Cell Injection Targeting GPRC5D OriCAR-017 in Patients With Relapsed and/or Refractory Multiplemyeloma
Brief Title: OriCAR-017 Chimeric Antigen Receptor (CAR) Modified T Cells for the Treatment of R/RMM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OriCell Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OriCAR-017-P1
Record Dates: First submitted 2023-12-11; First posted 2023-12-27 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-04

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OriCAR-017 ( GPCRC5D-directed chimeric antigen receptor modified T cells ) (Experimental): Phase I (Dose-Escalation) The subjects enrolled will be sequentially assigned to the corresponding dose level to determin the RP2D. The dose-escalation part of the study will adopt the the standard 3+3 design, wherein 3 dose levels are planned to be evaluated.
  Phase I (Dose-Expansion) After determining the RP2D, one of the dose levels will be selected for further evaluation during the dose-expansion part. Up to 10 to 15 additional subjects who are diagnosed with relapsed/refractory MM will be enrolled to further explore the anti-tumor activity of Ori-CAR-017.
  Phase II The Phase II part of the study will be initiated at the RP2D of OriCAR-017 which will be selected based on the clinical data obtained during the Phase I part of the study.
  Interventions: Biological: OriCAR-017

INTERVENTIONS:
Biological: OriCAR-017 — GPCRC5D-directed chimeric antigen receptor modified T cells

SUMMARY:
An open label, dose exploratory clinical study to evaluate the safety, efficacy, and pharmacokinetics of OriCAR-017 in R/RMM

DETAILED DESCRIPTION:
This is a Phase I and Phase II, open-label, multi-center study to assess the safety, pharmacokinetics, and efficacy of GPRC5D directed chimeric antigen receptor modified T cells injection (OriCAR-017) in n patients with relapsed and/or refractory multiplemyeloma (R/RMM).

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of R/RMM according to the IMWG criteria;
* Expected survival period is >12 weeks;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 or 2 at the time of ICF signature;
* The expression of GPRC5D in bone marrow plasma cells membrane is more than 20% by flow cytometry and/or immunohistochemistry, multiple myeloma with measurable lesions, and at least one of the following criteria must be met:

  1. Serum M protein >5 g/L;
  2. Urine M protein level >200 mg/24 hour;
  3. Serum free light chain (sFLC) >100 mg/L and K/λ FLC ratio is abnormal;
  4. Primitive immature or monoclonal plasma cells >5% by bone marrow cytology or flow cytometry.
* Subjects who had received at least 3 prior lines of therapy including (but not limited to) immunomodulatory drugs (IMiDs), proteasome inhibitors, anti-CD38 monoclonal antibodies, etc., but have failed treatment, including those who have experienced relapse (within 12 months), refractory or intolerant to the last line treatment regimen.

Main Exclusion Criteria:

* Smoldering myeloma (asymptomatic)
* Multiple myeloma with only extramedullary lesions;
* Plasma cell leukemia;
* Concurrent amyloidosis;
* Central nervous system metastasis, leptomeningeal disease or metastatic central compression;
* HBsAg or HbcAb is positive, and the quantitative detection of hepatitis B virus (HBV) DNA in peripheral blood is more than 100 copies/L; hepatitis C virus (HCV) antibody and HCV RNA in peripheral blood is positive; human immunodeficiency virus (HIV) antibody positive; syphilis antibody is positive at Screening; Cytomegalovirus DNA test is positive;
* Had hypersensitivity or intolerance to any drug/excipient (including conditioning chemotherapy) used in this study;
* Previously received treatment targeting GPRC5D, including but not limited to antibodies, ADC, or CAR-T;
* Subjects who received autologous hematopoietic stem cell transplantation (ASCT) within 8 weeks of Screening Visit or who plan to undergo ASCT during the study;
* Any uncontrolled active infection within 4 weeks prior to ICF signing or leukapheresis requires parenteral antibiotic, antiviral, or antifungal treatment
* Major surgery within 28 days prior to Screening Visit with the exception of a biopsy and an insertion of a central venous catheter or during the study;
* Subjects who received allogeneic stem cell therapy;
* Subjects complications or other conditions evaluated by investigators may affect compliance with the protocol or make them unsuitable to participate in this study;
* Pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-75
Enrollment: 83 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of OriCAR-017-P1 | Up to 28 days
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level.
Dose-limiting toxicity (DLT) | Up to 28 days
  tolerability

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until the date of first documented progression or date of death from any cause or withdraw, whichever came first, assessed up to 2 Years
  Objective response is defined as the participants with a partial response (PR) or better by the RECIST1.1 criteria.
Pharmacokinetics (the number of cell copies and cell persistence duration in peripheral blood) | From date of randomization until the date of first documented progression or date of death from any cause or withdraw, whichever came first, assessed up to 2 years
  CAR-GPRC5D DNA in peripheral blood detected by q-PCR at each visit after infusion
Antitumor efficacy-Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression
Antitumor efficacy-Duration of response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The period from the first evaluation of sCR or CR or VGPR or PR or MR to the first evaluation of PD or death of any cause
Long term survival follow up | From date of randomization until the date of first documented date of death from any cause, assessed up to 15 years
  The period from randomization until the date of death

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital College of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Beijing GoBroad Hospital, Beijing
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - Tongji Hospital of Tongji University, Shanghai
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No